CLINICAL TRIAL: NCT05916183
Title: Impact of Dehydration and Rapid Rehydration on Cognitive Function
Brief Title: Dehydration Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Riana Pryor, Assistant Professor, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007342
Record Dates: First submitted 2023-06-05; First posted 2023-06-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration | interventions — Economics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dehydration and Rehydration Arm (Experimental): Participants will complete exercise until 5% body mass loss, followed by ad libitum rehydration throughout 2 hours of recovery.
  Interventions: Behavioral: Fluid loss and consumption

INTERVENTIONS:
Behavioral: Fluid loss and consumption — Upon 5% body mass loss, rehydration of fluid lost to sweating throughout a 2 hour recovery period

SUMMARY:
The investigators want to understand the impact of the body losing and gaining water on brain function. Participants will restrict fluids consumed and exercise to lose 5% of body mass. Participants will then be provided fluid equal to the volume lost to consume over 2 hours (recovery). A series of brain function tests will be performed at baseline, following weight loss, and following recovery.

DETAILED DESCRIPTION:
A baseline series of brain function tests will be performed. Following this, participants will complete a 24 hour fluid and water rich food restriction on the day proceeding testing. Participants will then complete moderate to high intensity exercise in a hot/humid room to achieve 5% body mass loss. Once baseline core body temperature returns to baseline levels, the series of brain function tests will be performed. Participants will then consume a sports drink equal to the volume of sweat lost over the course of a 2 hour recover period. Following this, he series of brain function tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Recreationally active
* 18-26 years old

Exclusion Criteria:

* History of cardiovascular, metabolic, respiratory, neural, or renal disease
* Hypertensive (systolic blood pressure ≥ 140 mmHg, diastolic blood pressure ≥ 90 mmHg) or tachycardic (resting heart rate ≥ 100 bpm) during the screening visit
* Taking medication or supplements with a known side effect of affecting physiological responses to exercise (e.g., aspirin, acetaminophen, beta blockers, statins, stimulants, depressants, SSRIs)
* Tobacco or nicotine use in the past six months
* Current or past musculoskeletal injury impacting physical activity
* Study physician discretion based on any other medical condition or medication

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Multitasking test | Upon completion of 5% body mass loss protocol, approximately 2 hours into the trial
  Accuracy score of a multitasking test (0-100%) with greater scores indicating a better outcome
Multitasking test | 2 hours following the dehydration cognitive function test, approximately 4.5 hours into the trial
  Accuracy score of a multitasking test (0-100%) with greater scores indicating a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Riana R Pryor, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Coded data or the methodology will be shared with researchers upon reasonable written request.
Supporting Information: Study Protocol
Time Frame: Data can be shared for as long as the data is retained, at least 7 years.
Access Criteria: Data will be shared upon reasonable written request.